CLINICAL TRIAL: NCT03100617
Title: Single Arm Study of Modified REACH-VA Alzheimer's Caregiver Intervention in Vietnam
Brief Title: Alzheimer's Family Caregiver Intervention in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1084736
Record Dates: First submitted 2017-03-24; First posted 2017-04-04 (Actual); Results first posted 2020-03-16 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Dementia Alzheimers
Keywords: Family caregiver
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REACH-VA family caregiver intervention (Experimental): Behavioral intervention with several components including 1) caregiver education, 2) risk assessment, 3) caregiver needs assessment, 4) caregiver skill building and problem solving, and 4) caregiver stress reduction.
  Interventions: Behavioral: Psychosocial caregiver intervention

INTERVENTIONS:
Behavioral: Psychosocial caregiver intervention — Modified version of the REACH-VA intervention for family caregivers of persons with dementia. The intervention has several components including 1) caregiver education, 2) risk assessment, 3) caregiver needs assessment, 4) caregiver skill building and problem solving, and 4) caregiver stress reduction.

SUMMARY:
This is a single arm pilot study of 6-8 families to test the feasibility and acceptability of a Alzheimer's family caregiver intervention in Vietnam.

DETAILED DESCRIPTION:
This is a single arm pilot study of 6-8 families to test the feasibility and acceptability of a modified version of the REACH-VA caregiver intervention in Vietnam. The REACH-VA caregiver intervention is an evidence-based intervention that has been shown to be effective in multicultural populations in the US. The model has been modified for use in Vietnam. This study will test the modified model in Vietnam. Participants in this study will be adult family caregivers of non-institutionalized persons with dementia who are living in Hanoi, Vietnam. They will receive 4-6 sessions delivered over the course of 2-3 months that will included the following components: 1) education about the nature of the disease, 2) risk assessment, 3) enhancing caregiver skills and problem-solving, and 4) caregiver stress reduction. The intervention will be delivered by a social worker or nurse using a Vietnamese language versions of the REACH-VA protocol and caregiver intervention notebook.

ELIGIBILITY:
Inclusion Criteria:

* Primary adult family caregiver of person with dementia

Exclusion Criteria:

* Caregivers of persons with dementia who are institutionalized

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-26 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam National Geriatric Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: This group received the REACH-VA intervention
Period: Overall Study
Arm/Group | Treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | REACH-VA Family Caregiver Intervention
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 51.7 [43 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Vietnam | 6
Zarit Burden Scale 4-item [Mean (Full Range); unit: units on a scale] — This instrument measures the amount of caregiving burden experienced by the participant. Each of the 4 items on the Zarit Burden Inventory is rated from 0 (no burden) to 4 (high burden). The range is therefore from 0 (lowest level of burden) to 16 (highest level of burden).
  units on a scale | 7.8 [0 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Burden
Description: Zarit Burden scale
Time Frame: Change from baseline Zarit burden scale score to 3 months.
Population: This was a feasibility study. Outcome data not collected.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Treatment: Behavioral intervention
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
This was a small case series to examine acceptability and feasibility of the intervention and no outcome data were collected from the 6 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT03100617/Prot_000.pdf